CLINICAL TRIAL: NCT01917994
Title: Seek Test Treat Retain Strategies Leveraging Mobile Health Technologies
Brief Title: Text Messaging Intervention to Improve Retention in Care and Virologic Suppression in an Urban HIV-Infected Population
Acronym: Connect4Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA032057 (NIH)
Record Dates: First submitted 2013-08-01; First posted 2013-08-07 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: HIV; Patient Adherence; Mobile Technology
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text Messages + Appointment Reminders (Experimental): Participants in the intervention arm will receive supportive, informational, or motivational text messages three times a week for one year in addition to text message reminders about HIV primary care appointments.
  Interventions: Behavioral: Text Messages; Behavioral: Appointment Reminders
- Appointment Reminders (Active Comparator): Participants in the control arm will receive text messages reminding them of HIV primary care appointments 48 hours before the scheduled appointment.
  Interventions: Behavioral: Appointment Reminders

INTERVENTIONS:
Behavioral: Text Messages — The intervention consists of supportive, informational, and motivational text messages three times a week targeting the following domains: promoting a sense of connectedness to the clinic, fostering social support, building empowerment, ameliorating negative affect, cultivating positive affect, and promoting healthy behaviors and adherence to antiretroviral medication.
  Arms: Text Messages + Appointment Reminders
Behavioral: Appointment Reminders

SUMMARY:
Retention in care and virologic suppression are the key final steps of the HIV treatment cascade. Poor or intermittent retention has been associated with later initiation of antiretroviral therapy, virologic failure, and death. Regular HIV care has also been associated with a decrease in HIV transmission risk behavior. Despite the proven health and prevention benefits of consistent HIV care, only 40-50% of those infected with HIV in the United States are estimated to meet current retention in care standards and even fewer - only about 25% - are estimated to be virologically suppressed.

The Behavioral Model for Vulnerable Populations provides a useful framework for understanding broad areas that may impact adherence to care and treatment. Individual-level domains include vulnerable (e.g., depression, stigma), enabling (e.g., social support, positive affect), and need (e.g., co-morbidities) factors, and structural domains include, for example, features or the clinic and the provider-patient relationship.

Short message service (SMS) technology represents a new and exciting tool to help retain HIV-infected patients in care and treatment. SMS interventions have been deployed successfully in support of antiretroviral adherence and virologic suppression in sub-Saharan Africa, where two randomized trials have showed clear benefits. A pilot study conducted in our clinic suggests that use of SMS messages to promote adherence to care and treatment in the urban HIV-infected poor is both feasible and acceptable.

The investigators believe that combining SMS technology with content-specific messages designed to impact factors highlighted in the Behavioral Model for Vulnerable Populations can improve retention in care and virologic suppression for an urban public hospital population living with HIV, thus the investigators propose the following specific aims.

Specific Aim 1: Determine whether a behavioral theory-based SMS intervention improves virologic suppression [primary outcome] and retention in care [secondary outcome] for a vulnerable urban HIV-infected population through a randomized trial of this technology compared to SMS appointment reminders alone. Retention in care will also be analyzed as a mediator of virologic suppression. Exploratory outcomes include time to virologic suppression, sustained virologic suppression, emergency department utilization and antiretroviral adherence, as well as levels of depression, positive affect, social support and empowerment.

Specific Aim 2: Examine patient experiences with the SMS intervention, focusing specifically on: 1) satisfaction with this technology; 2) identifying barriers to and facilitators of patient use of this technology, and; 3) the preferred frequency and content of intervention messages.

Specific Aim 3: Conduct cost and cost-effectiveness analyses of the SMS intervention.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Age 18 or over
* English-speaking
* Able to give informed consent
* Have a cell phone and willing to send/receive up to 25 text messages/month
* Detectable viral load plus either 1) new to clinic (no more than 2 primary care visits) or 2) history of poor retention (one missed visit or lack of six-month visit constancy in the past year)

Exclusion Criteria:

* HIV-uninfected
* Under age 18
* Monolingual speaker of a language other than English
* Unable to give informed consent
* Undetectable viral load
* Perfect appointment adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Viral Load | 12 month

SECONDARY OUTCOMES:
Missed Visit Proportion | 12 month
  Number of missed or "no show" visits divided by number of scheduled appointments
Appointment Adherence | 12 month
  Each participant's proportion of kept appts divided by scheduled appts (mean of the proportions)
Visit Constancy | 12 month
  At least one kept visit in each six-month period
Attended All Scheduled Visits | 12 month
  Attended all scheduled visits

OTHER OUTCOMES:
Time to Virologic Suppression | 12 month
Sustained virologic suppression | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Christopoulos, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital Positive Health Program, San Francisco, California, United States

REFERENCES:
- [Background] Christopoulos KA, Riley ED, Tulsky J, Carrico AW, Moskowitz JT, Wilson L, Coffin LS, Falahati V, Akerley J, Hilton JF. A text messaging intervention to improve retention in care and virologic suppression in a U.S. urban safety-net HIV clinic: study protocol for the Connect4Care (C4C) randomized controlled trial. BMC Infect Dis. 2014 Dec 31;14:718. doi: 10.1186/s12879-014-0718-6. PMID 25551175
- [Derived] Christopoulos KA, Riley ED, Carrico AW, Tulsky J, Moskowitz JT, Dilworth S, Coffin LS, Wilson L, Johnson-Peretz J, Hilton JF. A Randomized Controlled Trial of a Text Messaging Intervention to Promote Virologic Suppression and Retention in Care in an Urban Safety-Net Human Immunodeficiency Virus Clinic: The Connect4Care Trial. Clin Infect Dis. 2018 Aug 16;67(5):751-759. doi: 10.1093/cid/ciy156. PMID 29474546